CLINICAL TRIAL: NCT05197413
Title: Study to Evaluate the Efficacy of Arrae's Bloat & Calm Alchemy Capsules to Reduce Bloating, Heartburn and Gas, and Alleviate the Intensity of IBS Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arrae (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20219Arrae
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: IBS - Irritable Bowel Syndrome; Anxiety
MeSH Terms: conditions — Irritable Bowel Syndrome; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arrae Bloat supplement (Experimental): The "Bloat" capsules are a blend of 5 herbs and a fruit-based digestive enzyme that target the cause for IBS symptoms.
  Interventions: Dietary Supplement: Arrae bloat supplement

INTERVENTIONS:
Dietary Supplement: Arrae bloat supplement — The supplement contains organic dandelion root extract, organic lemon balm herb top extract, organic peppermint leaf extract, organic bromelain, organic slippery elm inner bark extract. The capsule itself is made of cellulose, which is not a main active ingredient.

SUMMARY:
This is an open-label observational crossover trial to study the efficacy of a commercial dietary supplement and its effect on common symptoms of IBS (such as bloating, gas, heartburn, and other symptoms).

DETAILED DESCRIPTION:
It is hypothesized that the dietary supplement marketed as "Arrae Bloat" will improve subjective wellbeing in trial participants. It is further hypothesized that a second dietary supplement marketed as "Arrae Calm" will support the effects of "Arrae Bloat", while reducing stress, anxiety and panic and promoting restful sleep and easing tension in the body, which has previously been reported in customer feedback studies.

ELIGIBILITY:
Inclusion Criteria:

* Female over 18 years old
* Self-reported (undiagnosed) IBS symptoms, such as self-reported abdominal pain, gas production and bloating after meals, heartburn after meals
* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Following a stable, consistent diet regimen
* Agree to refrain from any lifestyle changes that may affect their GI tract and IBS symptoms for the duration of the study
* May have self-reported sleep issues
* May have self-reported mild anxiety/depression
* May have self-reported occasional panic attacks

Exclusion Criteria:

* Prior prescriptions for IBS
* Current IBS treatment (e.g. proton pump inhibitors, laxatives)
* Follow an extreme diet intervention
* Experienced severe weight loss in the past 3 months prior to study participation
* Antibiotic usage within 3 months prior of study participation
* Usage any medication or herbal remedies which can affect the GI tract
* Food intolerances/allergies
* Pineapple sensitivity/allergy
* Taking cortisol lowering prescription medication
* Has any of the following medical conditions:

History of GI tract cancers Celiac disease / gluten intolerance GI bleeding Rectal bleeding Heme-positive stool Iron-deficiency anemia Systemic signs of infection Insomnia Moderate to severe depression/anxiety Moderate to severe panic attacks

- Females that are pregnant, want to become pregnant for the duration of the study, or who are breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in IBS symptoms (bloating, heartburn and gas) | 4 weeks
  Survey-based assessment (0-5 scale with 0 being the lowest possible score and 5 being the highest) of changes in IBS symptoms between baseline and study intervention period.
Reduction in anxiety symptoms | 8 weeks
  Survey-based assessment (0-5 scale with 0 being the lowest possible score and 5 being the highest) of changes in anxiety symptoms between baseline and study intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No